CLINICAL TRIAL: NCT04835623
Title: Effects of CEQUA™ on Objective and Subjective Dry Eye Findings Associated With Sjogren's Syndrome
Brief Title: CEQUA for Sjogren's Syndrome Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Center for Ophthalmic and Vision Research, LLC (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-001
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Dry Eye; Dry Eye Syndromes; Sjogren's Syndrome
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome | interventions — Cyclosporine; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclosporine (Experimental): Participants receive Cyclosporine 0.09% Ophthalmic Solution (Cequa), 1 drop, each eye, twice a day for 12 weeks
  Interventions: Drug: Cyclosporine 0.09% Ophthalmic Solution

INTERVENTIONS:
Drug: Cyclosporine 0.09% Ophthalmic Solution — one drop each eye twice daily
  Other Names: Cequa Ophthalmic Product

SUMMARY:
The primary objective of this study is to show that CEQUA (cyclosporine 0.09% ophthalmic solution) improves symptoms of dry eye disease in a population of patients with Sjogren's Syndrome diagnosis.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving informed consent will have an eye exam and will be asked about their medical history to determine eligibility for the study. Eligible participants will continue to the second visit the same day or up to 10 days later. During the second visit participants will answer questionnaires about their eyes and have their vision, eyes, and tears examined. All participants will be given CEQUA to use over the duration of the study. The same procedures will be repeated every four weeks for 3 months total.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Sjogren's Syndrome.
* Self-reported complaints of ocular dryness for a period of at least 3 months
* Best-corrected distance visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

* Use of cyclosporine within the last 3 months.
* Use of ocular steroid within the 3 months.
* Previous history of treatment failure with cyclosporine.
* Known hypersensitivity or contraindication to the study medication or any of its ingredients.
* Use of any systemic or topical ocular medication that is known to cause or exacerbate dry eye.
* Any active ocular infection.
* Severe or serious ocular condition in either eye or any other unstable medical condition that may preclude study treatment or follow-up.
* History or presence of chronic generalized systemic disease that might increase the risk to the subject or confound the results of the study.
* Currently pregnant or lactating.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in total corneal staining | Baseline and week 12
  Expanded NEI corneal staining scale ranging from 0 to 15

SECONDARY OUTCOMES:
Mean change from baseline in total conjunctival staining | Baseline and week 12
  Expanded NEI conjunctival staining scale ranging from 0 to 20
Mean change from baseline in the score of dry eye questionnaires | Baseline and week 12
  Dry eye questionnaire score ranging from 0 to 28

CONTACTS AND LOCATIONS:
Overall Officials: John Rocco Robilotto, OD, PhD, Principal Investigator — Center for Ophthalmic and Vision Research
Locations (1):
- Center for Ophthalmic and Vision Recearch, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: No